CLINICAL TRIAL: NCT01650181
Title: Biochemical and Echosonographic Impacts Using Siliphos-Selenium-Methionine-Alpha Lipoic Acid + Metformin Versus Metformin in Patients With Fatty Liver and Steatohepatitis
Brief Title: Effects of Siliphos-Selenium-Methionine-Alpha Lipoic Acid in Patients With Fatty Liver and Non-alcoholic Steatohepatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, M.D. Science Master, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GAS-399-11/11/1
Record Dates: First submitted 2012-07-11; First posted 2012-07-26 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Liver Disease
Keywords: nafld, nash, fatty liver
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Metformin; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Patients treated with diet, exercise and metformin
  Interventions: Drug: Metformin
- Suplement (Active Comparator): Patients treated with diet, exercise and metformin plus Siliphos (140mg) + Selenium (15mcg) -Methionine 3mg + Alpha Lipoic Acid (200mg).
  Interventions: Dietary Supplement: Siliphos+ Selenium - Methionine + Alpha Lipoic Acid

INTERVENTIONS:
Drug: Metformin — Patients with Steatohepatitis treated with diet, exercise and metformin
  Arms: Metformin
Dietary Supplement: Siliphos+ Selenium - Methionine + Alpha Lipoic Acid — Patients with Steatohepatitis treated with diet, exercise, metformin and Siliphos (140mg) + Selenium (15 mcg) - Methionine (3mg) + Alpha Lipoic Acid (200mg), two tablets BID
  Arms: Suplement
Dietary Supplement: Siliphos+ Selenium - Methionine + Alpha Lipoic Acid — Patients with fatty liver treated with diet, exercise, metformin and Siliphos (140mg) + Selenium (15 mcg) - Methionine (3mg) + Alpha Lipoic Acid (200mg), two tablets BID
  Arms: Suplement
Drug: Metformin — Patients with fatty liver treated with diet, exercise and metformin
  Arms: Metformin

SUMMARY:
Non-alcoholic steatohepatitis represents 10 - 15% total cases of hepatic cirrhosis. In the upcoming years, the economic burden of this disease will increase and will mean an important problem for our health system due to obesity epidemic.

There are several treatments for non-alcoholic steatohepatitis; however, none of them have overcome a healthy lifestyle including diet, exercise and some drugs related with insulin metabolism.

There after, using hepatoprotective drugs and antioxidants have been recommended as an eligible therapy to reduce the progression from fatty liver to steatohepatitis and cirrhosis. Being this approach not only an experimental item yet but also an unavoidable reality.

The purpose of this randomized controlled study is explore the effects of siliphos-selenium-methionine-alpha lipoic acid + metformin versus metformin in patients with fatty liver and non-alcoholic steatohepatitis about biochemical and echosonographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Metabolic Syndrome according to ATP III Criteria
* Non smokers
* Without intake of vitamins or herbal medicine for at least one month
* Without uncontrolled glycemic levels
* Compatible ultrasound and/or histological report

Exclusion Criteria:

* Alcohol ingest > 50 gr weekly or chronic alcoholism
* Creatine serum > 2 mg/dL
* Potassium serum > 5.5 mEq/L
* Allergic to metformin or any components of the study
* Pregnancy
* Anomalies of blood coagulation or liver anatomic
* Patients with diseases and/or treatment that cause fatty liver or steatohepatitis
* Body weight change > 10% in the last 5 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Impact on biochemical and echosonographic parameters | 6 months
  Identify and measure if patients with metabolic syndrome with NALFD under Siliphos (140mg) + Selenium (15mcg) - Methionine (3mg) + Alfa lipoic acid (200mg) treatment added to conventional therapy improves echosonographic pattern measure accord bright scale and biochemical parameters like LFT´s compared with conventional therapy alone (metformin + diet + exercise).

SECONDARY OUTCOMES:
Identify changes in anthropometric parameters | 6 months
  Identify and measure changes in anthropometrics parameters of metabolic syndrome like BMI, fasting glucose, lipid profile, arterial pressure, abdominal perimeter, waist index.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, M.D., M. Sc., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico